CLINICAL TRIAL: NCT05428033
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Determine the Efficacy and Safety of Once Daily Centanafadine Capsules for the Treatment of Children With Attention-deficit/Hyperactivity Disorder (ADHD)
Brief Title: A Trial of Centanafadine Efficacy and Safety in Children With Attention-deficit/ Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405-201-00021
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Attention Deficit/Hyperactivity Disorder
Keywords: Centanafadine; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 1-(naphthalen-2-yl)-3-azabicyclo(3.1.0)hexane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Weight Based High Dose Centanafadine Capsules (Experimental): Cohort 1, (6 to 12 years of age)
  Cohort 2, (4 to 5 years of age)
  High dose - weight-based dosing
  Interventions: Drug: centanafadine capsule
- Weight Based Low Dose Centanafadine Capsules (Experimental): Cohort 1, (6 to 12 years of age)
  Low dose - weight-based dosing
  Interventions: Drug: centanafadine capsule
- Matching Placebo (Placebo Comparator): Cohort 1 and Cohort 2
  Children (4 to 12 years of age, inclusive) to receive Placebo capsules will be matching in size and color.
  Interventions: Other: placebo capsule

INTERVENTIONS:
Drug: centanafadine capsule — capsule
  Other Names: centanafadine; centanafadine XR; EB-1020
  Arms: Weight Based High Dose Centanafadine Capsules; Weight Based Low Dose Centanafadine Capsules
Other: placebo capsule — capsule
  Other Names: placebo comparator; matching placebo
  Arms: Matching Placebo

SUMMARY:
This trial will be conducted to evaluate the efficacy of centanafadine QD XR versus placebo in the treatment of child subjects (4 to 12 years, inclusive) with ADHD. The trial will consist of a screening period, a double-blind treatment period, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 4 to 12 years (inclusive) at the time of informed consent/assent.
* A primary diagnosis of ADHD based on DSM-5 diagnosis criteria as confirmed with the MINI-KID.
* A minimum symptoms total raw score of ≥ 28 on the ADHD-RS-5 at baseline for all subjects.
* A score of 4 or higher on the CGI-S-ADHD at baseline.
* Subjects aged 4 or 5 years only: has failed adequate psychotherapy or in the investigator's opinion, is severe enough to require pharmacotherapy in the absence of prior psychotherapy.

Exclusion Criteria:

* Comorbid diagnosis of: Tourette's Disorder, Generalized Anxiety Disorder that is severe enough to interfere with trial procedures, Panic Disorder, Conduct Disorder, Psychosis, Post-traumatic Stress Disorder, Bipolar Disorder, Autism Spectrum Disorder, Oppositional Defiant Disorder that is severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), Obsessive-Compulsive Disorder that is severe enough to interfere with trial conduct (allowed if it is not the primary focus of treatment), or MDD with current major depressive episode.
* A significant risk of committing suicide based on history and the investigator's clinical judgment, or routine psychiatric status examination, Current suicidal behavior, Imminent risk of injury to self, Active suicidal ideation. A history of suicidal behavior (over the last 6 months).
* BMI ≥ 40 kg/m2 or ≤ 5th percentile for age and gender based on US CDC criteria.
* Has initiated, changed, or discontinued receiving psychological interventions for ADHD within the 30 days before the screening visit, or is anticipated to start new treatment during the trial.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 574 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Attention-Deficit/Hyperactivity Disorder Rating Scale Version 5 (ADHD-RS-5) Change from baseline in the ADHD-RS-5 symptoms total raw score (investigator interview with informant) at Week 6 | From baseline to week 6

SECONDARY OUTCOMES:
Clinical Global Impression - Severity - Attention-Deficit/Hyperactivity Disorder (CGI-S-ADHD) change from baseline in CGI-S-ADHD at Week 6 | From baseline to week 6
Conners-3 Parent Short- Change from baseline in Conners-3 Parent Short at Week 6 | From baseline to week 6

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com